CLINICAL TRIAL: NCT06992934
Title: Non Interventional Study Aiming to Assess the Immunological Impact of a Post Cell Therapy Treatment With FLT3 Inhibitors on the Phenotype, the Metabolism, the Function of T-cells and Monocytes and Macrophages
Brief Title: Immunological Impact of a Post Cell Therapy Treatment With FLT3 Inhibitors
Acronym: TARGETALLO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-AOI-11
Record Dates: First submitted 2025-04-22; First posted 2025-05-28 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gilteritinib (Experimental): Administration of Gliteritinib
  Interventions: Drug: Gilteritinib

INTERVENTIONS:
Drug: Gilteritinib — Administration of Gilteritinib

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (aHSCT) is the only curative option for many hematological maligancies. The main cause of death following HSCT is the relapse of the original disease.

Few strategies have been developed to prevent relapse after bone marrow transplantation. New prophylactic strategies are needed to decrease the relapse incidence without increasing the non-relapse mortality in the post-transplant area. Several drugs are currently being explored as maintenance in several AML subgroups such as FLT3 ITD/mutated AML.

A specific group of AML patients display the FMS-like tyrosine kinase 3 (FLT3) internal tandem duplication (ITD) or mutation. These recurrent genetic abnormalities account for 30-35% of all AML patients. Because FLT3 is a tyrosine kinase, it can be targeted using tyrosine kinase inhibitors (TKI). Originally limited to first generation sorafenib and Midostaurin, the FLT3 TKI now include second generation Gilteritinib, crenolanib and quizartinib13. Because many FLT3 AML patients would relapse after aHSCT, the use of sorafenib, the only FLT3 TKI available at that time, in a post-transplant setting started to be evaluated.

Sorafenib is a multi-kinase inhibitor that not only inhibit FLT3 but also the RAS, RAF, KIT, and the VEGF and platelet-derived growth factor receptor. Several retrospective trials reported the safety and efficiency of a sorafenib maintenance.

In recent years, a mounting piece of evidence suggests that sorafenib may have an impact on several immune cells as T cell populations, dendritic cells, macrophages and myeloid-derived immunosuppressor cells (MDSC). Other more potent and more specific FLT3 inhibitors are currently under investigation both in combination with chemotherapy before transplantation and as post transplantation maintenance. In this line, crenolanib and Gilteritinib are two potent and more specific TKI that proved more effective than sorafenib in the treatment of FLT3 ITD/TKD relapsed, refractory AML patients. These drugs demonstrated a higher response rate in R/R patients. These two drugs are part of the future standard of care in FLT3 AML but their immunological impact has never been studied.

At a time where cellular therapies (allogeneic stem cell transplantation but also CAR T cells) and targeted therapies are becoming the central point of cancer treatment, it appears mandatory to better understand the interactions between the two. The goal of our research project which covers fundamental and clinical aspects of AML post-transplant treatments is devoted to a better understanding of the impact of Gilteritinib on the immune cells in order to rationalize their use after aHSCT. A better characterization of the action of these drugs on the immune system is urgently needed to develop new prophylactic strategies which could decrease the relapse incidence without increasing the non-relapse mortality in the post-transplant area. This program is proposed for a period of 3 years, time necessary to perform all the in vitro and ex vivo approaches and to recruit a sufficient number of patients eligible for aHSCT.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18y/o
* Patient who received an allogeneic stem cell transplantation for an acute myeloid leukemia and who will receive gilteritinib as post transplantation maintenance
* Matched related, matched unrelated, mismatched unrelated and haploidentical donors

Exclusion Criteria:

* Minors
* Pregnant women
* Patient under 'tutelle', 'curatelle' or in prison
* Patient who has been treated for a solid tumor in the past 2 years
* Known human immunodeficiency virus (HIV) infection or HIV-related malignancy
* Clinically active hepatitis B or hepatitis C infection
* Known allergy or hypersensitivity to gilteritinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Assess the off-target effects of Gilteritinib on the phenotype of immunity cells | At 3 months, 6 months, 1 year post maintenance start
  Evaluation of the phenotype
Assess the off-target effects of Gilteritinib on the function of immunity cells | At 3 months, 6 months, 1 year post maintenance start
  Evaluation of the phenotype
Assess the off-target effects of Gilteritinib on the metabolism of immunity cells | At 3 months, 6 months, 1 year post maintenance start
  Evaluation of the phenotype

SECONDARY OUTCOMES:
Overall survival after transplant | At 3 months post-transplant, 6 months, 1-year post
  record of survival status
transplant relapse free survival | At 3 months post-transplant, 6 months, 1-year post
  record of relapse event
aGVHD incidence | At 3 months post-transplant, 6 months, 1-year post
  record of aGVHD event
cGVHD incidence | At 3 months post-transplant, 6 months, 1-year post
  record of cGVHD event
Infection incidence | At 3 months post-transplant, 6 months, 1-year post
  record of infection event

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
Not planned